CLINICAL TRIAL: NCT02780089
Title: A US Multi-Site Observational Study in Patients With Unresectable And Metastatic Melanoma: The OPTIMIzE Study
Brief Title: Study in Patients With Unresectable And Metastatic Melanoma: The Optimize Study
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-357
Record Dates: First submitted 2016-04-25; First posted 2016-05-23 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Melanoma
Keywords: Metastatic; Unresectable
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- Prospective Patients: There will be 1,600 prospective patients recruited over a period of two years and followed-up for a planned minimum of three years. For the prospective cohort, patients will be recruited after the course of treatment has been decided by the physician and prior to the start of treatment.Prior advanced melanoma treatment information will be collected from patient charts for pre-treated patients. Patients will be followed for a minimum of 3 years from their study index date until death, withdrawal of consent, lost to follow-up/record, or end of study, whichever comes first. Study index date will be the date when first study therapy is initiated.
- Treatment Group No. 1: Immune checkpoint inhibitor patients who remain on an immune checkpoint inhibitor therapy. Defined as immune checkpoint inhibitor therapy patients who either remained on their initial (index) immune checkpoint inhibitor therapy or switched to another immune checkpoint inhibitor therapy during the study period. Patients in this group remained on an immune checkpoint inhibitor therapy and did not switch to a non-immune checkpoint inhibitor therapy anytime during the study period.
- Treatment Group No. 2: Immune checkpoint inhibitor patients who switched to a non-immune checkpoint inhibitor therapy. Defined as patients who switched from their index immune checkpoint inhibitor therapy to a non-immune checkpoint inhibitor therapy anytime during the study period.
- Treatment Group No. 3: Targeted therapy patients who remain on a targeted therapy. Defined as targeted therapy patients who either remained on their initial (index) targeted therapy or switched to another targeted therapy during the study period. Patients in this group remained on a targeted therapy and did not switch to a non-targeted therapy anytime during the study period.
- Treatment Group No. 4: Targeted therapy patients who switched to a non-targeted therapy. Defined as patients who switched from their index targeted therapy to a non-targeted therapy anytime during the study period.
- Treatment Group No. 5: Chemotherapy/other therapy patients who remain on a chemotherapy/other therapy. Defined as chemotherapy/other therapy patients who either remained on their initial (index) chemotherapy/other therapy or switched to another chemotherapy/other therapy during the study period. Patients in this group remained on a chemotherapy/other therapy and did not switch to an immune checkpoint inhibitor therapy or targeted therapy anytime during the study period.
- Treatment Group No. 6: Chemotherapy/other patients who switched to an immune checkpoint inhibitor therapy or targeted therapy. Defined as patients who switched from their index chemotherapy/other therapy to an immune checkpoint inhibitor therapy or targeted therapy anytime during the study period.
- Retrospective Patients: Retrospective cohort of 600 patients with unresectable or metastatic melanoma, receiving therapies other than immune checkpoint inhibitor or targeted therapies during the four year period prior to the release of ipilimumab (March 25, 2007 -March 24, 2011), will be identified. The data for these 600 retrospective patients will be used as a benchmark for treatment patterns and outcomes prior to the marketed availability of immune checkpoint inhibitors or targeted therapies.

SUMMARY:
This study evaluates the different patterns of care for patients who have unresectable or metastatic melanoma. The dosing, duration, regimen, indication, and treatments will be observed. The survival rate of these patients will also be observed.

DETAILED DESCRIPTION:
This is a non-interventional, observational study with the primary objective to assess and describe "real world" patterns of care in the treatment of patients with unresectable or metastatic melanoma. A sample size of 1,600 prospective patients will provide sufficient information to explore this primary objective. There will be no forced number of patients enrolled into a specific treatment cohort. Setting or controlling specific treatment enrollment cohort counts would invalidate the results of the primary objective of the study. No primary hypothesis is being tested.

ELIGIBILITY:
Inclusion Criteria:

Prospective cohort patients:

* Diagnosis date must occur on or after March 24, 2011 (date of ipilimumab approval in US)
* Diagnosis of stage III (unresectable) or stage IV melanoma (includes mucosal, uveal acral-lentiginous, leptomeningeal disease)
* Age ≥ 18 years at time of entry into study
* Patients must be actively receiving or scheduled to receive systemic treatment (any line, eg, first, second, third line [including investigational drugs]).

  * For patients initiating new treatment, treatment must be started within 28 days after signing informed consent.
  * For patients currently receiving treatment, patients must enroll within the first 21 days of starting new treatment

Retrospective cohort patients:

* Patients with diagnosis of confirmed unresectable stage III or stage IV melanoma (including mucosal, uveal, acral-lentiginous, leptomeningeal disease)
* Age ≥ 18 years at time of unresectable or metastatic melanoma diagnosis
* Initiated therapy for unresectable or metastatic melanoma within 4 years prior to approval of ipilimumab (first immune checkpoint inhibitor therapy approved in US)

  * March 25, 2007 - March 24, 2011
* One year of follow-up data is required from date of therapy initiation, if a patient passed away within the one year of follow-up; such patients are still eligible and the date of death will be collected.

  1. If retrospective patients have at least one year of follow-up data and are then treated with immuno-oncology, immune checkpoint inhibitor therapy, or targeted therapy, these patients will be analyzed separately.

Exclusion Criteria:

Prospective patients:

* Patients participating in a clinical study that does not allow enrollment into a non interventional study or clinical studies in which the investigational treatment is blinded
* Patients who started new treatment > 21 days
* Patients who enrolled in study but did not initiate treatment before 28 days
* Patients with current malignancies (except non-melanoma skin cancer and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) that requires additional systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with histologically-confirmed unresectable stage III or stage IV melanoma, (including mucosal, uveal, acral-lentiginous, leptomeningeal disease). Patients can be treatment-naïve or previously treated for unresectable or metastatic melanoma.
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Patterns of Care | Up to 5 years
  To assess the selection and sequencing of drugs and practice patterns used to treat unresectable and metastatic melanoma (e.g. immune checkpoint agents, targeted agents, or combination therapies) in a real-world setting. Reasons for initial treatment decisions across and between drug classes, changes in treatment, and discontinuation will be recorded (e.g. lack of benefit, safety, cost, or other barriers to care).
Demographics | Up to 5 years
  Baseline characteristics (age, gender, race/ethnicity)
Overall Survival | Up to 5 years
  To estimate overall survival in patients receiving therapy for unresectable or metastatic melanoma some statistical measurements and actual survival will be used.
Disease Characteristics | Up to 5 years
  Disease characteristics (date of diagnosis, disease stage, performance status)

SECONDARY OUTCOMES:
Healthcare Resource | up to 5 years
  To compare and describe healthcare utilization, imputed costs, and impact of initial treatment choice on lifetime or periodic costs. Due to potential differences between in patterns of care among various regions, region-specific analyses may be conducted for healthcare resource utilization.
Functional Assessments of Cancer Therapy-Melanoma (FACT-M) | Up to 12 months
European Quality of Life-5 Dimensions (EQ-5D) | Up to 12 months
Work Productivity and Activity Impairment: General Health (WPAI:GH) | Up to 12 months
The Caregiver Quality of Life Index - Cancer (CQOLC) | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (66):
- United States (66):
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Pacific Shores Medical Group, Long Beach, California
  - Cancer Care Associates, Redondo Beach, California
  - University of Colorado, Aurora, Colorado
  - 21st Century Oncology, Jacksonville, Florida
  - Cancer Specialits, LLC D/B/A, Jacksonville, Florida
  - Lakeland Regional Health, Lakeland, Florida
  - Watson Clinical Center for Research, INC, Lakeland, Florida
  - UF Health Cancer Center at Orlando Health, Longwood, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Mid Florida Hematology and Oncology Centers, Orange City, Florida
  - Sacred Heart Medical Oncology Group, Pensacola, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center Moffitt Cancer Center, Tampa, Florida
  - Harbin Clinic, Rome, Georgia
  - Summit Cancer Care, Savannah, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - North Shore University Health System, Evanston, Illinois
  - Ingalls Cancer Research Center, Harvey, Illinois
  - Oncology Specialits, S.C., Niles, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Simmons Cancer Institute at SIU School of Medicine, Springfield, Illinois
  - Stormont-Vail Cancer Center, Topeka, Kansas
  - University of Kansas Medical Center, Westwood, Kansas
  - West Ky Hematology & Oncology, Paducah, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - CHRISTUS Schumpert Cancer Treatment Center, Shreveport, Louisiana
  - Saint Agnes Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center (MCCC), Rochester, Minnesota
  - Forrest General Cancer Center, Hattiesburg, Mississippi
  - Central Care Cancer Center, Bolivar, Missouri
  - Nebraska Hematology-Oncology, P.C., Lincoln, Nebraska
  - Oncology Hematology West P.C., Omaha, Nebraska
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Atlantic Health, Morristown Medical Center, Morristown, New Jersey
  - Meridian Health, Neptune City, New Jersey
  - Rosewell Park Cancer Institute, Buffalo, New York
  - Center of Learning Healthcare, Durham, North Carolina
  - Hematolgoy and Oncology Associates, Inc., Canton, Ohio
  - Aultman Hospital, Canton, Ohio
  - Tri-County Hematology and Oncology Associates, Inc, Massillon, Ohio
  - Genesis Cancer Care Center, Zanesville, Ohio
  - St. Charles Medical Center - Cancer Center, Bend, Oregon
  - Network Office of Research & Innovation / Lehigh Valley Health Network, Allentown, Pennsylvania
  - St. Luke's Hospital and Health Network, Bethlehem, Pennsylvania
  - The Regional Cancer Center, Erie, Pennsylvania
  - Lancaster General Health, Lancaster, Pennsylvania
  - Jefferson Medical Oncology, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - UPCI - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Texas Oncology, Austin, Texas
  - Texas Oncology, El Paso, Texas
  - Texas Oncology, Paris, Texas
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah
  - Inova Melanoma and Skin Cancer Center, Fairfax, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - Cancer Care Northwest, Spokane, Washington
  - West Virginia University, Bridgeport, West Virginia
  - West Virginia University, Huntington, West Virginia
  - West Virginia University Hematolgoy & Oncology, Martinsburg, West Virginia
  - West Virginia University, Morgantown, West Virginia
  - Gundersen Lutheran Medical Foundations, Inc., La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kirkwood JM, Kottschade LA, McWilliams RR, Khushalani NI, Jang S, Hallmeyer S, McDermott DF, Tawbi H, Che M, Lee CH, Ritchings C, Le TK, Park B, Ramsey S. Real-world outcomes with immuno-oncology therapies in advanced melanoma: final results of the OPTIMIzE registry study. Immunotherapy. 2024 Jan;16(1):29-42. doi: 10.2217/imt-2022-0292. Epub 2023 Nov 8. PMID 37937397
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome